CLINICAL TRIAL: NCT01477983
Title: Kansai Plus Atrial Fibrillation Trial; UNmasking Dormant Electrical Reconduction by Adenosine TriPhosphate Trial; Efficacy of Antiarrhythmic Drugs Short-Term Use After Catheter Ablation for Atrial Fibrillation Trial
Brief Title: Kansai Plus Atrial Fibrillation Trial
Acronym: KPAF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kyoto University, Graduate School of Medicine (Other)
Responsible Party: Principal Investigator, Satoshi Shizuta, Satoshi Shizuta, Kyoto University, Graduate School of Medicine, Kyoto University, Graduate School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KPAFKUHP
Record Dates: First submitted 2011-11-12; First posted 2011-11-23 (Estimated); Last update posted 2017-08-18 (Actual); Status verified 2017-08

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; catheter ablation; adenosine triphosphate; antiarrhythmic drugs
MeSH Terms: conditions — Atrial Fibrillation | interventions — Anti-Arrhythmia Agents; Flecainide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- ATP guide additional ablation - AAD (Active Comparator): UNDER-ATP trial: ATP guide additional ablation, EAST-AF trial: AAD for 90 days
  Interventions: Procedure: ATP guide additional ablation.; Drug: Antiarrhythmic drug (AAD)
- Control - AAD (Active Comparator): UNDER-ATP trial: Control, EAST-AF trial: AAD for 90 days
  Interventions: Procedure: Control; Drug: Antiarrhythmic drug (AAD)
- ATP guide additinal ablation - Control (Active Comparator): UNDER-ATP trial: ATP guide additional ablation, EAST-AF trial: Control
  Interventions: Procedure: ATP guide additional ablation.; Drug: Control
- Control - Control (Active Comparator): UNDER-ATP trial: Control, EAST-AF trial: Control
  Interventions: Procedure: Control; Drug: Control

INTERVENTIONS:
Procedure: ATP guide additional ablation. — Following successful PV isolation, intravenous ATP of 0.4 mg/body-weight-kg is rapidly is injected, and dormant LA-PV conduction is evaluated. If dormant LA-PV conduction is unmasked, then additional radiofrequency energy applications are delivered to the conduction gaps until disappearance of dormant LA-PV conduction.
  Other Names: The brand names of ATP; Adetphos-L, Trinosin-S
  Arms: ATP guide additional ablation - AAD
Drug: Antiarrhythmic drug (AAD) — Following successful ablation, AAD (Vaughan Williams class I or III) is administered for 90 days. The recommended drugs are flecainide, propafenone, sotalol and amiodarone, but the final choice of drug and dosage is left to the discretion of the attending physician.
  Other Names: Brand names; Tambocor, Pronon, Sotacor, Ancaron
  Arms: ATP guide additional ablation - AAD
Procedure: ATP guide additional ablation. — Following successful PV isolation, intravenous ATP of 0.4 mg/body-weight-kg is rapidly is injected, and dormant LA-PV conduction is evaluated. If dormant LA-PV conduction is unmasked, then additional radiofrequency energy applications are delivered to the conduction gaps until disappearance of dormant LA-PV conduction.
  Other Names: The brand names of ATP; Adetphos-L, Trinosin-S
  Arms: ATP guide additinal ablation - Control
Drug: Control — Following successful ablation, AAD (Vaughan Williams class I or III) including flecainide, propafenone, sotalol and amiodarone is not used during the period of 0 - 90 days.
  Other Names: Brand names; Tambocor, Pronon, Sotacor, Ancaron
  Arms: ATP guide additinal ablation - Control
Procedure: Control — Following successful PV isolation, intravenous ATP is not administered.
  Other Names: The brand names of ATP; Adetphos-L, Trinosin-S
  Arms: Control - AAD
Drug: Antiarrhythmic drug (AAD) — Following successful ablation, AAD (Vaughan Williams class I or III) is administered for 90 days. The recommended drugs are flecainide, propafenone, sotalol and amiodarone, but the final choice of drug and dosage is left to the discretion of the attending physician.
  Other Names: Brand names; Tambocor, Pronon, Sotacor, Ancaron
  Arms: Control - AAD
Procedure: Control — Following successful PV isolation, intravenous ATP is not administered.
  Other Names: The brand names of ATP; Adetphos-L, Trinosin-S
  Arms: Control - Control
Drug: Control — Following successful ablation, AAD (Vaughan Williams class I or III) including flecainide, propafenone, sotalol and amiodarone is not used during the period of 0 - 90 days.
  Other Names: Brand names; Tambocor, Pronon, Sotacor, Ancaron
  Arms: Control - Control

SUMMARY:
This is a 2x2 factorial randomized controlled trial (KPAF Trial), evaluating two different pharmacological approaches to improve long-term outcome of catheter ablation for atrial fibrillation (AF). The study is composed of UNmasking Dormant Electrical Reconduction by Adenosine TriPhosphate (UNDER-ATP) Trial and Efficacy of Antiarrhythmic Drugs Short-Term Use after Catheter Ablation for Atrial Fibrillation (EAST-AF) Trial. Patients with paroxysmal or persistent AF will be randomized to ATP guide ablation or control group in a 1:1 ratio before the procedure (UNDER-ATP Trial). Excluding those with severe procedural complications or substantial bradycardia identified first after ablation for persistent AF, patients will be randomized in a 1:1 ratio to antiarrhythmic-drug (AAD) or control group after the procedure (EAST-AF Trial).

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is a common tachyarrhythmia causing disabling symptoms and stroke. Although catheter ablation has been developed as curative therapy for AF, it is still associated with considerably high rate of AF recurrence, approximately 30-40% in patients with paroxysmal AF and 50-80% among those with persistent AF.

Because most ectopic beats triggering AF originate from myocardial sleeves in pulmonary veins (PVs), the mainstay of catheter ablation for AF is PV isolation. The major cause of early and late AF recurrence following successful PV isolation is considered to be electrical reconnection between left atrium (LA) and PVs. Therefore, it is important to establish permanent LA-PV disconnection, although high energy application is associated with increased risk of procedural complications, including cardiac tamponade, PV stenosis/occlusion and LA-esophageal fistula.

Adenosine or adenosine triphosphate (ATP) has been reported to unmask dormant electrical conduction between LA and PVs after successful PV isolation. Thus, adenosine or ATP guide additional ablation until disappearance of dormant electrical conduction has been proposed as adjunctive approach to establish permanent LA-PV disconnection and thereby decrease AF recurrence post ablation. However, only several small observational studies showed the efficacy of adenosine or ATP guide ablation, and this approach is not recognized as standard therapy.

On the other hand, sizable portion of AF recurrence early after ablation is considered to be due to irritability in LA from the ablation. Thus, short term use of antiarrhythmic drugs (AADs) after ablation has been proposed as adjunctive approach not only to prevent early AF recurrence, but also to improve long-term outcome by promoting reverse remodeling of LA through maintenance of sinus rhythm during the first 2-3 months period after ablation.

The 5A study, a recently reported single-center study, randomized 110 patients with paroxysmal AF to AAD or control group. In the AAD group, AAD was used for 6 weeks after ablation. Although AAD significantly reduced early AF recurrence during the first 6 weeks, discontinuation of the drug resulted in similar AF-free rates at 6 months. Considering the small number of patients enrolled in the 5A study, the results were not conclusive, lacking statistical power to determine the effect of short-tem use of AAD following successful ablation for AF on long-term clinical outcome. Also, this approach is expected to be more effective in patients with persistent AF rather than those with 'self-terminating' paroxysmal AF. In addition, 6 weeks may have been too short to promote reverse remodeling of LA.

Accordingly, we planned a 2x2 factorial randomized controlled trial (KPAF trial), evaluating the efficacy of ATP guide additional ablation and 90 days use of AADs post ablation. Approximately 2,000 patients with paroxysmal or persistent AF will be randomized to ATP guide ablation or control group in a 1:1 ratio before the procedure (UNDER-ATP trial). Excluding those with severe procedural complications or those with substantial bradycardia identified first after ablation for persistent AF, patients will be randomized in a 1:1 ratio to AAD or control group after the procedure (EAST-AF trial). Approximately 5% of the patients are expected to be excluded from the EAST-AF trial after ablation, but those patients will not be excluded from the UNDER-ATP trial, whose data will be analyzed by intention-to-treat manner. The follow-up duration is one year.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing first catheter ablation including PV isolation for paroxysmal or persistent atrial fibrillation
* Patients who are 21-79 years old
* Able to be followed for one year in an out-patient clinic
* Willing to sign the consent form for participation

Exclusion Criteria:

* Contraindication or intolerance to adenosine triphosphate or Vaughan Williams class I or III antiarrhythmic drugs, including severe bronchial asthma, severe vasospastic angina, and substantial bradycardia including sinus node dysfunction with prolonged pauses on termination of atrial fibrillation
* Age =< 20 years or => 80 years
* Renal insufficiency (serum creatinine >=2.0mg/dl or hemodialysis)
* NYHA class IV heart failure
* Left ventricular ejection fraction < 40%
* Left atrial diameter > 55mm
* Very long-lasting (>=5years) persistent atrial fibrillation
* Ineligible for optimal anticoagulant therapy
* History of myocardial infarction within the past 6 months
* Prior or planned open heart surgery
* Severe valve heart disease
* Unable to be followed in an out-patient clinic for one year
* Unwilling to sign the consent form for participation
* When the attending physician are unwilling to enroll the patient in the study
* When the attending physician consider inappropriate to enroll the patient in the study
* Those with severe procedural complications (EAST-AF trial only)

Ages: 21 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2113 (Actual)
Dates: Start 2011-11; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Atrial tachyarrhythmias lasting for > 30 seconds or requiring repeat ablation, hospital admission, cardioversion or antiarrhythmic drug (AAD) therapy between 91 and 365 days after ablation. (Both trials) | 91 - 365 days
  Atrial tachyarrhythmias include atrial fibrillation, atrial tachycardia, and common or uncommon atrial flutter.
  Antiarrhythmic drug (AAD) indicates Vaughan Williams class I or III drug.

SECONDARY OUTCOMES:
Repeat Ablation for atrial tachyarrhythmias. (Both trials) | 0 - 365 days
Atrial tachyarrhythmias lasting for > 30 seconds or requiring repeat ablation, hospital admission, cardioversion or antiarrhythmic drug (AAD) therapy* between 0 and 90 days after ablation. (Both trials) | 0 - 90 days
  * In patients assigned to AAD group, AAD therapy between 0 and 90 days post ablation is not regarded as this secondary outcome.
Atrial tachyarrhythmias lasting for > 30 seconds or requiring repeat ablation, hospital admission, cardioversion or antiarrhythmic drug (AAD) therapy* after ablation. (Both trials) | 0 - 365 days
  * In patients assigned to AAD group, AAD therapy between 0 and 90 days post ablation is not regarded as this secondary outcome.
Quality of Life (QOL) score. (Both trials) | 0 - 365 days
  Atrial Fibrillation Quality of Life Questionnaire（AFQLQ) is used in this study.
Procedural complications including cardiac tamponade, thromboembolism, PV stenosis/occlusion, left atrium-esophageal fistula, and peri-esophageal injury. (UNDER-ATP trial) | 0 - 365 days
Total procedure time. (UNDER-ATP trial) | Day-0
Total fluoroscopy time. (UNDER-ATP trial) | Day-0
Total radiation dose. (UNDER-ATP trial) | Day-0
Total number and duration of radiofrequency energy applications. (UNDER-ATP trial) | Day-0
Total number and duration of radiofrequency energy applications for pulmonary vein isolation. (UNDER-ATP trial) | Day-0
Side effects of ATP including bronchial asthma, angina and sustained hypotension (<90mmHg or requiring vasopressor) during and after the procedure. (UNDER-ATP trial) | 0 - 365 days
Side effects of antiarrhythmic drugs (EAST-AF trial) | 0 - 365 days

CONTACTS AND LOCATIONS:
Overall Officials: Satoshi Shizuta, MD, Principal Investigator — Department of Cardiovascular Medicine, Kyoto University Graduate School of Medicine
Locations (1):
- Division of Cardiology, Kyoto University Hospital, Kyoto, Japan